CLINICAL TRIAL: NCT00525707
Title: Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel Group Study to Assess the Efficacy, Safety, and Tolerability of Tezosentan in Patients With Acute Heart Failure.
Brief Title: Tezosentan in Acute Heart Failure
Acronym: VERITAS 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-051-306
Record Dates: First submitted 2007-08-31; First posted 2007-09-06 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Acute Heart Failure; Acute Decompensation of Chronic Heart Failure; New Onset of Heart Failure
Keywords: acute heart failure; Actelion; tezosentan; acute decompensation of chronic heart failure; New onset of heart failure
MeSH Terms: interventions — tezosentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): tezosentan delivered i.v. at 20 mL/h (5 mg/h) for 30 min followed by 4ML/h (1 mg/h) for 23.5 to 71.5 h (24 to 72 h in total)
  Interventions: Drug: tezosentan
- 2 (Placebo Comparator)
  Interventions: Drug: tezosentan

INTERVENTIONS:
Drug: tezosentan — tezosentan delivered i.v. at 20 mL/h (5 mg/h) for 30 min followed by 4ML/h (1 mg/h) for 23.5 to 71.5 h (24 to 72 h in total)

SUMMARY:
The randomized patients with acute heart failure will be stratified based on the presence or absence of a Swan-Ganz catheter and assigned to receive either tezosentan 5 mg/h for the first 30 minutes and 1 mg/h thereafter or matching placebo in a 1:1 manner. The duration of the treatment is 24 hours up to 72 hours. The duration of the follow-up period is 30 days after treatment initiation for death, re-hospitalizations and SAEs followed by a follow-up period of 5 months for vital status.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older.
2. Male or non-breast-feeding, non-pregnant female (only females who are post menopausal, surgically sterile or practicing a reliable method of contraception).
3. Acute heart failure (ischemic or non-ischemic).
4. Randomization within 24 hours of hospitalization (including emergency room stay) for acute heart failure.
5. Dyspnea at rest as assessed by the patient and breathing rate ³ 24/min (measured during 60 seconds).
6. At least two out of the following four criteria: · elevated BNP or N terminal pro-BNP (more than three times the upper limit of normal for the site) in patients not treated with nesiritide,· clinical evidence of pulmonary congestion/edema (e.g., rales or crackles more than a third above bases),· evidence of pulmonary congestion on chest X-ray, · left ventricular systolic dysfunction (EF < 40% or wall motion index £ 1.2 within 12 months prior to randomization).
7. Patients in need of i.v. therapy for acute heart failure and who have received at least one dose of i.v. diuretic within 24 hours prior to study drug initiation (last bolus dose must have been more than 2 hours prior to study drug initiation).
8. Written informed consent.

Exclusion Criteria:

Criteria only for patients hemodynamically monitored:

1. Baseline cardiac index > 2.5 l/min/m2 and/or PCWP < 20 mmHg within 6 hours prior to study drug initiation.

   Criteria for all patients:
2. Patients not receiving i.v. vasodilators (e.g., nitrates, nitroprusside, nesiritide) at baseline: supine systolic blood pressure < 100 mmHg. Patients receiving i.v. vasodilators (e.g., nitrates, nitroprusside, nesiritide) at baseline: supine systolic blood pressure < 120 mmHg.
3. Cardiogenic shock within the last 48 hours or evidence of volume depletion.
4. Ongoing myocardial ischaemia, coronary revascularisation procedure (PCI or CABG) during current admission or planned revascularisation.
5. ST-segment elevation myocardial infarction or administration of thrombolytic therapy.
6. Baseline creatinine ≥ 2.5 mg/dl (221 mmol/l).
7. Baseline hemoglobin < 10 g/dl or a hematocrit < 30%.
8. Hemodialysis, ultrafiltration or peritoneal dialysis within the last 7 days.
9. Heart failure due to active myocarditis, obstructive hypertrophic cardiomyopathy, congenital heart disease, restrictive cardiomyopathy or constrictive pericarditis. Heart failure caused by valvular disease.
10. Acute heart failure associated with uncontrolled hemodynamically relevant atrial fibrillation/flutter or ventricular rhythm disturbances.
11. Acute heart failure secondary to clinical evidence of digoxin toxicity or any other drug-related toxicity.
12. Significant chronic and/or acute lung disease that might interfere with the ability to interpret the dyspnea assessments or hemodynamic measurements (e.g., severe chronic obstructive pulmonary disease or acute pneumonia).
13. Mechanical circulatory or ventilatory support. Prior CPAP use is allowed, if discontinued at least 2 hours prior to study drug initiation.
14. Acute systemic infection/sepsis or other illness with a life expectancy less than 30 days.
15. Coronary artery bypass graft, or other cardiac surgery, or major non-cardiac surgery within the last 30 days.
16. Patients who received another investigational drug within 30 days prior to randomization.
17. Re-randomization in the current study.
18. Any factors that might interfere with the study conduct or interpretation of the results such as known drug or alcohol dependence.
19. Concomitant treatment with cyclosporin A or tacrolimus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 735 (Actual)
Dates: Start 2003-04; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Incidence of death or worsening heart failure | 7 days following study drug initiation

SECONDARY OUTCOMES:
effect on patient's dyspnea assessment, measured using a visual analog scale | Over first 24 hours

CONTACTS AND LOCATIONS:
Locations (35):
- United States (8):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - Advanced Heart Failure and Transplant Service, Palo Alto VA Health Care System, Cardiology Section, Palo Alto, California
  - Denver VAMC, Denver, Colorado
  - The Heart Hospital at Alledgheny General, Division of Cardiology, Pittsburgh, Pennsylvania
  - Veterans Affairs Medical Center, Houston, Texas
  - Tyler Cardiovascular Consultants, Tyler, Texas
  - Danville Medical Center, Danville, Virginia
  - Medical Associates, Bellebue, Bellevue, Washington
- AKH University of Vienna, Abt. Medizinische Kardiologie, Vienna, Austria
- Roskilde Amt Sygehus, Roskilde, Denmark
- France (4):
  - Hopital Ambroise Pare, Service de Cardiologie, Boulogne
  - Heart Failure clinic C.H. Dubos, Pontoise
  - Hopitaux Universitaires de Strasbourg, Hopital Hautepierre, Strasbourg
  - CHU Rangueil, Cardiologie A, Toulouse
- Germany (3):
  - Medizinische Klinik I, Universitatsklinikum Aachen, Aachen
  - Campus Virchow-Klinikum, Medizinishe Klinik mit Schwerpunkt Kardiologie, Berlin
  - Georg-August-Universitat Gottingen, Zentrum fur Innere Med, Göttingen
- Dept. of Cardiology, University of Athens, Alexandra Hospital, Athens, Greece
- Israel (6):
  - Barzilai Hospital, Ashkelon
  - Carmel Medical Center, Haifa
  - Wolfson Medical Center, Holon
  - Hadassah Hospital, Jerusalem
  - Nazareth Hospital EMMS, Nazareth
  - Assaf-Harofeh Medical Center, Ẕerifin
- Poland (5):
  - Klinika Kardiologii i Chorob Wewnetrznych, Samodzielny Publiczny Szpital, Bydgoszcz
  - Klinika Chorob Serca, Akademia Medyczna w Gdansku, Gdansk
  - I Klinika Kardiolgii, Collegium Medicum UJ, Krakow
  - Institute of Cardiology College, College of Medicine of Jagellonian University, Krakow
  - Kategra I Klinika Kardiolgii AM, Wroclaw
- Switzerland (3):
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne
  - Cardio Centro Ticino, Servizio Cardiovasculare, Lugano
  - University Hospital Zurich, Zurich
- United Kingdom (3):
  - Glasgow Royal Infirmary, Glasgow
  - Hull Royal Infirmary, Hull
  - Scunthorpe General Hospital, Scunthorpe

REFERENCES:
- [Derived] Cotter G, Davison BA, Milo O, Bourge RC, Cleland JG, Jondeau G, Krum H, O'Connor CM, Metra M, Parker JD, Torre-Amione G, van Veldhuisen DJ, Kobrin I, Rainisio M, Senger S, Edwards C, McMurray JJ, Teerlink JR; VERITAS Investigators. Predictors and Associations With Outcomes of Length of Hospital Stay in Patients With Acute Heart Failure: Results From VERITAS. J Card Fail. 2016 Oct;22(10):815-22. doi: 10.1016/j.cardfail.2015.12.017. Epub 2015 Dec 22. PMID 26721775
- [Derived] McMurray JJ, Teerlink JR, Cotter G, Bourge RC, Cleland JG, Jondeau G, Krum H, Metra M, O'Connor CM, Parker JD, Torre-Amione G, van Veldhuisen DJ, Lewsey J, Frey A, Rainisio M, Kobrin I; VERITAS Investigators. Effects of tezosentan on symptoms and clinical outcomes in patients with acute heart failure: the VERITAS randomized controlled trials. JAMA. 2007 Nov 7;298(17):2009-19. doi: 10.1001/jama.298.17.2009. PMID 17986694